CLINICAL TRIAL: NCT01287598
Title: A Phase I, Non-randomized Open-label Study to Evaluate the Effect of BAY73-4506 (Regorafenib) on Probe Substrates of CYP 2C9 (Warfarin), 2C19 (Omeprazole) and 3A4 (Midazolam) in a Cocktail Approach (Group A) and on a Probe Substrate of CYP 2C8 (Rosiglitazone, Group B) in Patients With Advanced Solid Tumors
Brief Title: BAY73-4506 Probe Substrate Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12434
Record Dates: First submitted 2011-01-31; First posted 2011-02-01 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Neoplasms
Keywords: Phase I; Probe substrate; target therapy; small molecule; pharmacokinetics
MeSH Terms: conditions — Neoplasms | interventions — regorafenib; Warfarin; Omeprazole; Midazolam; Rosiglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Regorafenib (Stivarga, BAY73-4506) + warfarin + omeprazole + midazolam
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506); Drug: Warfarin; Drug: Omeprazole; Drug: Midazolam
- Arm 2 (Experimental): Regorafenib (Stivarga, BAY73-4506) + rosiglitazone
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506); Drug: Rosiglitazone

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — BAY73-4506 administered once a daily (od) in a 21-day on / 7-day off schedule
Drug: Warfarin — CYP 2C9 (warfarin) at Cycle 1
  Arms: Arm 1
Drug: Omeprazole — CYP 2C19 (omeprazole) at Cycle 1
  Arms: Arm 1
Drug: Midazolam — CYP 3A4 (midazolam) at Cycle 1
  Arms: Arm 1
Drug: Rosiglitazone — CYP2C8 (rosiglitazone) at Cycle 1
  Arms: Arm 2

SUMMARY:
* To evaluate the effect of BAY73-4506 on the pharmacokinetics of probe substrates of CYP 2C9 (warfarin), 2C19 (omeprazole) and 3A4 (midazolam) administered in a cocktail approach and on the pharmacokinetics of a probe substrate of CYP 2C8 (rosiglitazone)
* To evaluate safety, anti-tumor activity, pharmacokinetics, and pharmacodynamics of BAY73-4506 in patients with advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects must be ≥ 18 years at the first screening examination / visit
* ECOG Performance Status of ≤ 2
* Histological or cytological documentation of confirmed advanced solid tumors. Subjects should have measurable or non-measurable disease according to RECIST
* Life Expectancy of at least 3 months
* Adequate bone marrow, liver, and renal functions as assessed by the following laboratory requirements conducted within 14 days prior to the first study treatment:

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥1,500/mm3
  * Platelet count ≥ 100,000/ mm3
  * Total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
  * Alkaline phosphatase ≤ 2 times ULN
  * ALT and AST ≤ 2.5 x ULN (≤ 5.0 x ULN for subjects with cancer involving the liver)
  * Serum creatinine ≤ 1.5 times ULN and glomerular filtration rate (GFR)≥ 30 ml/min/1.73 m2, according to the MDRD (Modified Diet in Renal Disease) abbreviated formula
  * Lipase ≤ 1.5 ULN
  * INR and PTT ≤ 1.5 ULN
* Subjects who are therapeutically treated with warfarin, heparin or other anticoagulants are not eligible for study participation in Group A. Subjects who are therapeutically treated with warfarin, heparin or other anticoagulants, will be allowed to participate in Group B of the study provided they meet all eligibility criteria. Close monitoring of at least weekly evaluations will be performed until INR or PTT are stable by the local standard of care.
* Recovery from previous drug/procedure-related toxicities to CTC Grade 0 or 1 levels (except for alopecia), or to baseline preceding the prior treatment. Preexisting chemotherapy induced sensory neuropathy of CTC Grade ≤2 is not an exclusion criteria.
* Negative serum pregnancy test must be obtained within 7 days prior to the start of treatment in women of childbearing potential. Negative results must be available prior to study treatment.
* Subjects enrolled in this study must use adequate barrier birth control measures prior to, during the course of the study, and 3 months after the last administration of regorafenib.
* An adequate contraception includes the use of condoms or a vasectomy, hormonal contraception with implants or combined PO contraceptives, certain intrauterine devices, bilateral tubal ligation, or hysterectomy. In addition, adequate birth control measures for the subject's partner is required, such as a hormonal contraception with implants or combined PO contraceptives, certain intrauterine devices, bilateral tubal ligation, or hysterectomy, use of condoms or a vasectomy.

Exclusion Criteria:

* History of cardiac disease: Congestive heart failure (New York Heart Association, NYHA, Class III or IV) or active coronary artery disease (unstable angina [angina symptoms at rest] or new-onset angina [began within the last 3 months] or myocardial infarction within the past 6 months). Treatment with Type 1A or 3 anti-arrhythmics, such as Quinidine, Procainamide, Amiodarone, or Sotalol are not permitted. β-Blockers and digoxin are permitted.
* Left ventricular ejection fraction (LVEF) < 50% or below the LLN for the institution (whichever is higher).
* Subjects with pheochromocytoma
* Dehydration NCI-CTCAE, version 4, Grade > 1
* Uncontrolled hypertension (failure of diastolic blood pressure to fall to or below 90 mmHg or systolic blood pressure to fall to or below 140 mmHg with or without the use of antihypertensive drugs). At screening, subjects with history of hypertension should be on a stable anti-hypertensive treatment for at least 7 days prior to the first dose of study drug.
* Patients with known allergy to any of the study drug(s) to be administered, including known severe allergies, non-allergic drug reactions, or multiple drug allergies to any of the study drug(s) to be administered. This is also includes hypersensitivity to any of the compounds or excipients that will be administered to the study subject, specifically regorafenib, and warfarin, omeprazole and midazolam for subjects in Group A, or rosiglitazone for subjects in Group B.
* Subjects with arterial or venous thrombotic or embolic events, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, or pulmonary embolism within 6 months before the start of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-08-02 (Actual); Primary Completion 2018-07-03 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of probe substrates (AUC, Cmax, etc.) | Approximately 6 weeks

SECONDARY OUTCOMES:
Tumor Response evaluation measured by Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to 3 years or longer if indicated
Adverse event collection | Up to 3 years or longer if indicated

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (4):
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency-Vancouver Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec